CLINICAL TRIAL: NCT03162848
Title: Impact of SystemCHANGE™ Intervention on Medication Adherence in Older Adults With Heart Failure: A Pilot RCT
Brief Title: SystemCHANGE™ Intervention on Medication Adherence in Older Adults With Heart Failure
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Angela Andrews, PhD Student, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-130
Record Dates: First submitted 2017-05-11; First posted 2017-05-22 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Medication Adherence; Heart Failure; Aging
MeSH Terms: conditions — Medication Adherence; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SystemCHANGE intervention (Experimental): The SystemCHANGE™ intervention utilizes the Socioecological Model and Plan-Do-Check Act model as its framework and focuses on changing the individual's environment to change behavior using small experiments with feedback.
  Interventions: Behavioral: SystemCHANGE
- Attention Control (No Intervention): The attention control group will receive education at baseline, 1 month, and 2 months following America Heart Association brochures.

INTERVENTIONS:
Behavioral: SystemCHANGE — At initial home visit, the PI will work with the participant to identify important people for medication taking, routines, and cycles of routines. Possible solutions to incorporate medication taking into routines will be identified by the participant and PI and the participant will start implementing these solutions. Medication adherence will continuously be monitored using medication event monitoring systems. At one month, the participant will be sent a report on medication taking and a phone call will occur with the PI to discuss if solutions improved medication adherence or if other solutions need to be implemented. At month two, the intervention will end but participants are urged to continue to use solutions long term.
  Arms: SystemCHANGE intervention

SUMMARY:
The purpose of this pilot RCT study is to evaluate the acceptability and feasibility of a SystemCHANGE™ intervention to improve medication adherence in older adults with heart failure. The intervention focuses on changing the individual's environment by incorporating medication taking into existing routines using small experiments with feedback, and receiving support from people who impact routines.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years or older
* HF diagnosis confirmed by their physician utilizing their most recent ejection fraction
* prescribed diuretics
* self-administering medications
* able to open an electronic cap
* able to speak, hear and understand English
* not hospitalized,
* no cognitive impairment as determined by a score of 4 or greater on the 6-item mini-mental status exam.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility using open ended questionnaire | one point in time at the end of the maintenance phase which is 3 months after randomization into groups
  open ended questionnaire asking participants about acceptability and feasibility

SECONDARY OUTCOMES:
Systems thinking using questionnaire | baseline and after 2 month intervention phase
  questionnaire asking about personal systems behavior perceptions
Kansas City Cardiomyopathy Questionnaire | baseline and after 2 month intervention phase
  heart failure outcomes - SOB, fatigue, swelling, activity tolerance
Medication adherence using medication event monitoring systems | after randomization through end of maintenance phase for a total of 3 months
  Medication event monitoring systems

CONTACTS AND LOCATIONS:
Overall Officials: Angela Andrews, PhD(c), Principal Investigator — University of Missouri, Kansas City
Locations (1):
- Belleville Memorial, Belleville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No